CLINICAL TRIAL: NCT03328650
Title: Clinical Outcomes of the ALPS Proximal Humerus Plating System
Acronym: ALPS PHP
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Mihir Desai, Assistant Professor of Orthopaedic Surgery and Rehabilitation, Vanderbilt University Medical Center
Other Study IDs: 171043
Record Dates: First submitted 2017-10-09; First posted 2017-11-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Proximal Humeral Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Proximal Humerus Fracture Patients: As part of their routine care, patients who have experienced a proximal humerus fracture that requires operative fixation will receive the A.L.P.S® Proximal Humerus Plating System. This study is an observational, prospective study that monitors the patient's pain, functional ability, and patient-reported outcomes.

SUMMARY:
The purpose of this study is to document the performance and clinical outcomes of the A.L.P.S® Proximal Humerus Plating System.

Specific Aims:

* Conduct physical assessments measuring shoulder strength and range of motion, physician assessment of radiographs
* Obtain patient-reported outcomes regarding pain level, function capabilities, and work/leisure restrictions
* Document revisions, complications, and adverse events

DETAILED DESCRIPTION:
The purpose of this study is to document the performance and clinical outcomes of the A.L.P.S® Proximal Humerus Plating System.

Specific Aims:

* Conduct physical assessments measuring shoulder strength and range of motion, physician assessment of radiographs
* Obtain patient-reported outcomes regarding pain level, function capabilities, and work/leisure restrictions
* Document revisions, complications, and adverse events

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with a proximal humerus fracture requiring primary or revision ORIF using A.L.P.S Proximal Humerus Plating System
* Patients who present with a proximal humerus fracture that involves the metaphysis
* 18 years or older

Exclusion Criteria:

* Patients under the age of 18
* Patients who have an infection, sepsis, or osteomyelitis
* Patients who are unwilling to take part in study, have documented psychiatric disorder that limits ability to consent and maintain follow-up, or who may have severe problems maintaining follow-up (e.g. patients who are prisoners, homeless, intellectually changed without adequate family support)
* Patients who do not speak English (do to unavailability of non-English surveys)
* Patients who have known risk factors of pathologic fractures (e.g. bone metastasis)
* Patients who have received treatment for osteoporosis (e.g. bisphosphonate) within the last 5 years or whose treatment lasted longer than 5 years
* Patients who have Type 1 diabetes
* Patients who have other bone disease (e.g. osteogenesis imperfecta, Paget's disease, thyroid disease, Vitamin D deficiency, hyperparathyroidism)
* Patients that have a history of cancer, abnormal serum calcium, or chronic steroid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered a proximal humerus fracture that requires operative intervention using the A.L.P.S Proximal Humerus Plating System.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-08-07 (Actual); Primary Completion 2031-12-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone Material Strength | During surgical procedure
  Measured by the Osteoprobe
Bone Indentation Distance | During surgical procedure
  Measured by the Osteoprobe

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Orthopaedics, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available to other researchers.